CLINICAL TRIAL: NCT04486859
Title: A Prospective, Multicenter, Randomized Controlled Study of Postoperative Initiation of Thromboprophylaxis in Patients With Cushing's Disease
Brief Title: Postoperative Thrombosis Prevention in Patients With CD
Acronym: PIT-CD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Zhaoyun Zhang, vice director of endocrine department, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KY2020-794
Record Dates: First submitted 2020-07-22; First posted 2020-07-27 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Cushing Disease; DVT; Pulmonary Embolism
MeSH Terms: conditions — Pituitary ACTH Hypersecretion; Pulmonary Embolism

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mechanical prevention (Other): patients were managed with IPC
  Interventions: Device: IPC
- mechanical plus anticoagulant drugs prevention (Other): patients were managed with IPC, and LMWH was added 24h after surgery and followed by rivaroxaban 5 days after surgery
  Interventions: Drug: LMWH/Rivaroxaban; Device: IPC

INTERVENTIONS:
Drug: LMWH/Rivaroxaban — combined prevention
  Arms: mechanical plus anticoagulant drugs prevention
Device: IPC — mechanical prevention

SUMMARY:
Patients with Cushing disease was randomized to 2 groups. After surgery, the patients were managed with mechanical prevention or mechanical prevention plus anticoagulant drugs(LMWH followed by rivaroxaban), VTE was observed 24h, 5day, 4weeks and 12weeks after surgery.Bleeding events were also recorded.

DETAILED DESCRIPTION:
Cushing disease, caused by ACTH-secreting pituitary adenomas, can lead to serious complications with increased mortality. Minimally invasive surgery is currently the preferred treatment for the disease, allowing more than 80% of tumors to be completely removed. However, postoperative venous thrombosis (VTE), including deep vein thrombosis (DVT) and pulmonary embolism (PE) pose great threats to patients' safety. According to the literatures and the data from our center, up to 27% of the patients with Cushing's disease developed VTE after surgery. Due to the lacking of a randomized prospective study, there is no consensus or guideline on preventative anticoagulation protocols for postoperative management in patients with Cushing's disease. This is a prospective randomized control study on preventative anticoagulation in patients with Cushing's disease after transsphenoidal resection.

ELIGIBILITY:
Inclusion Criteria:

* Cushing's disease diagnosed and treated with transsphenoid surgery at study centers

Exclusion Criteria:

1. History of VTE before surgery or within 24 hours post-surgery
2. Acute bacterial endocarditis
3. Major bleeding events
4. Thrombocytopenia
5. Active gastrointestinal ulcers
6. History of stroke
7. High risk of bleeding due to clotting abnormalities
8. Participation in other clinical trials within the last three months
9. Contraindications to rivaroxaban (e.g., renal dysfunction with eGFR < 50 mL/min)
10. Presence of other malignant diseases
11. Severe mental or neurological disorders
12. Presence of intracranial vascular abnormalities
13. Contraindications to mechanical prophylactic anticoagulation
14. Pregnancy
15. Any other condition that researchers deem inappropriate for study participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
VTE incidence rate | 12 weeks
  DVT and PE incidence in 12 weeks after surgery

SECONDARY OUTCOMES:
DVT incidence rate | 12 weeks
  DVT in 12 weeks after surgery
PE incidence rate | 12 weeks
  PE in 12 weeks after surgery
Mortality | 12 weeks
  All-cause Mortality and VTE-specific Mortality
Symptomatic VTE incidence rate | 12 weeks
  Symptomatic DVT and PE incidence in 12 weeks after surgery

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - The First Affiliated Hospital of Sun Yat sen University, Guangzhou, Guangdong
  - Tongji Hospital, Wuhan, Hubei
  - Huashan Hospital, Shanghai, Shanghai Municipality
  - China West Hospital, Chengdu, Sichuan
  - People's Hopital of Xinjiang Uygur Autonomous Region, Ürümqi, Xinjiang
  - Peking Union Medical College Hospital, Beijing

REFERENCES:
- [Derived] Qiao N, He M, Ye Z, Gong W, Ma Z, Yu Y, Wu Z, Lu L, Zhu H, Yao Y, Liao Z, Wang H, Tan H, Cai B, Yu Y, Lei T, Yang Y, Jiang C, Yan X, Guo Y, Chen Y, Ye H, Wang Y, Tritos NA, Zhang Z, Zhao Y. Postoperative Initiation of Thromboprophylaxis in patients with Cushing's Disease (PIT-CD): a randomized controlled trial. Trials. 2025 Jun 21;26(1):217. doi: 10.1186/s13063-025-08923-6. PMID 40544300

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-06-12): https://cdn.clinicaltrials.gov/large-docs/59/NCT04486859/SAP_000.pdf